CLINICAL TRIAL: NCT02819804
Title: Phase Ib Study of Nivolumab and Dasatinib in Patients With Relapsed/Refractory Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia (Ph+ ALL)
Brief Title: Nivolumab and Dasatinib in Treating Patients With Relapsed or Refractory Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to funding and accrual issues
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 15H13; STU00202846 (CTRP (Clinical Trial Reporting Program)); NU 15H13 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-00711 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: B Acute Lymphoblastic Leukemia With t(9;22)(q34;q11.2); BCR-ABL1; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Refractory Adult Acute Lymphoblastic Leukemia; Refractory Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dasatinib, nivolumab) (Experimental): Patients receive dasatinib PO QD on days 1-28 and nivolumab IV over 30 minutes on days 8 and 22 of course 1 and on days 1 and 15 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacological Study

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Pharmacological Study — Correlative studies

SUMMARY:
The purpose of this research study is to determine the acceptable upper limit dose of nivolumab in combination with dasatinib that may be given to patients with relapsed/refractory philadelphia chromosome positive acute lymphoblastic leukemia (Ph+ ALL). Nivolumab is currently Food and Drug Administration (FDA) approved for other cancers, but has not yet been investigated in Ph+ ALL. Dasatinib is currently FDA approved for the treatment of Ph+ ALL, but has not yet been investigated in combination with nivolumab for this disease. There is evidence that dasatinib not only blocks the Philadelphia chromosome or breakpoint cluster region-Abelson murine leukemia viral oncogene homolog 1 (BCR-ABL) mutation, but also increases the activity of cells in your immune system. Nivolumab increases T cells in your immune system, which allows your immune system to attack the cancer. We think the combination of these drugs will be more effective against your leukemia than either drug used alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of nivolumab when given in combination with dasatinib in patients with relapsed/refractory Philadelphia chromosome positive (Ph+) acute lymphoblastic leukemia (ALL).

SECONDARY OBJECTIVES:

I. To evaluate the toxicities and safety profile of nivolumab and dasatinib in patients with relapsed/refractory Ph+ ALL.

II. To determine the rate of complete hematologic remission (CR) after three cycles of nivolumab and dasatinib.

III. To determine the rate of molecular remission after three cycles of nivolumab and dasatinib.

IV. To study the pharmacokinetics of nivolumab and dasatinib. V. To evaluate programmed cell death 1 (PD1) expression levels and saturation in the peripheral blood and bone marrow.

VI. To measure peripheral T-cell levels and activation in response to treatment.

TERTIARY OBJECTIVES:

I. To evaluate the 30 day mortality rate, overall survival (OS), progression free survival (PFS), and duration of remission (DOR) one year after treatment with nivolumab when given in combination with dasatinib in patients with relapsed/refractory Ph+ ALL.

II. To compare the OS between patients who receive a hematopoietic stem cell transplant and those who receive no further therapy following remission.

III. To evaluate for resistance mutations at the time of disease progression.

OUTLINE:

Patients receive dasatinib orally (PO) once daily (QD ) on days 1-28 and nivolumab intravenously (IV) over 30 minutes on days 8 and 22 of course 1 and on days 1 and 15 of subsequent courses. Courses repeat every 28 days in the absence of disease progression, unacceptable toxicity, or withdrawal from the study for other reasons.

After completion of study treatment, patients are followed up at 30 days and then monthly for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of Ph+ ALL
* Detection of one of the following must be present:

  * t(9;22)(q34;q11) or 3-way variant by metaphase cytogenetics
  * Breakpoint cluster region (BCR)-Abelson (ABL) positive status by molecular analysis with qualitative polymerase chain reaction (PCR) or fluorescence in situ hybridization (FISH)
* Patients must have primary refractory ALL based on failure to achieve a hematologic or molecular remission after induction therapy with dasatinib and steroids or dasatinib and chemotherapy, or have relapsed after treatment with a tyrosine kinase inhibitor with or without chemotherapy

  * Note: Prior course of dasatinib and steroid induction therapy should have included dasatinib 140mg PO daily on days 1-84 and prednisone 60mg/m^2 (capped at 120mg, or equivalent steroid dose) on days 1-28; if patients were unable to tolerate full steroid dose during induction therapy they will still be eligible
  * Note: Patients with refractory or relapsed disease in the central nervous system will be eligible
* Prior chemotherapy or tyrosine kinase inhibitor (TKI) treatment, aside from dasatinib, must be >= 7 days before first investigational agent dose
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must have adequate organ and bone marrow function prior to registration, as defined below:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2 x institutional upper limit of normal (IULN)
  * Total bilirubin < 2.0 x IULN (unless Gilbert syndrome has been diagnosed); if leukemia infiltration of the liver is suspected to be causing liver function abnormalities the patient will still be eligible with principal investigator (PI) approval
  * Creatinine < 2 x IULN
  * Creatinine clearance > 40 mL/min (measured by Cockroft-Gault)
* Females of child-bearing potential (FOCBP) must have a negative pregnancy test within 7 days of registration

  * Note: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Women must not be breastfeeding at the time of study registration
* Women and men of reproductive potential should agree to use two effective means of birth control

  * For women, contraception should continue for 23 weeks after the last dose of nivolumab and 12 weeks after the last dose of dasatinib to allow complete clearance of drug and its principal metabolites from the body
  * For men, contraception should continue for 31 weeks after nivolumab and 12 weeks after dasatinib
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients may not be receiving any other investigational agents within 5 half-lives of the drug (if known); if the half-life is not known, investigational agents should not be taken within two weeks
* Patients are not eligible if they have an intolerance to most recent prior TKI (other than dasatinib) at the lowest possible effective dose, defined as a grade >= 3 toxicity considered at least possibly related to that TKI; patients are also excluded if they are intolerant or allergic to dasatinib and discontinued prior therapy due to a >= grade 2 treatment related adverse event
* Patients must not have a history of a grade 4 anaphylactic reaction to monoclonal antibody therapy or known hypersensitivity reactions to drugs formulated with polysorbate 90
* Patients must not have had any prior therapy with an anti-PD-1, anti-programmed cell death 1 ligand 1 (PD-L1), anti-programmed cell death 1 ligand 2 (PD-L2), anti-cluster of differentiation (CD)137 or anti-cytotoxic t-lymphocyte-associated protein 4 ligand (CTLA-4) antibody (or any antibody or drug specifically targeting T-cell costimulation or checkpoint pathways; for questions or uncertainties, please contact the PI or quality assurance manager (QAM)
* Patients who have had allogeneic hematopoietic stem cell transplant (HSCT) are not eligible if they meet any of the following:

  * transplant is within 2 months from cycle 1, day 1 (C1D1)
  * Has clinically significant graft-versus-host disease requiring treatment
  * Has >= grade 3 persistent non-hematological toxicity related to the transplant
* Concomitant use of strong inhibitors of the cytochrome p450, family 3, subfamily a, polypeptide 4 (CYP3A4) isoenzyme is not permitted; must have wash-out period of 5 times the half-life of the compound before first dasatinib dose
* Concomitant use of QT prolonging agents strongly associated with torsades de pointes is not permitted
* Patients who have a known dasatinib-resistant ABL-kinase mutation such as T315I are not eligible; for confirmation, please contact PI
* Patients who have any serious or uncontrolled medical disorder that would impair the ability of the subject to receive protocol therapy are not eligible; these include, but are not limited to:

  * Active infection that is not well controlled
  * Known pleural or pericardial effusion at baseline
  * Clinically significant gastrointestinal disease or digestive dysfunction compromising absorption of dasatinib
  * Pulmonary arterial hypertension
  * Uncontrolled or significant cardiovascular disease, including:

    * Myocardial infarction within 6 months of enrollment date
    * Uncontrolled angina or congestive heart failure within 3 months of enrollment date
    * Left ventricular ejection fraction (LVEF) < 40%
    * Significant cardiac conduction abnormality, including:

      * History of clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
      * History of second or third degree heart block (except for second degree type 1)
      * Corrected QT (QTc) interval > 500 msec, unless a cardiac pacemaker is present
  * Prior malignancy active within the previous 3 years, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancers, superficial bladder cancer, or carcinoma in situ of the prostate, cervix or breast
  * Subjects with active, known or suspected autoimmune disease; (Note: Subjects with vitiligo, type I diabetes mellitus, hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll)
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing are not eligible
* Patients are not eligible if they have a known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (hepatitis C virus [HCV] antibody) indicating acute infection; Note: Patients with evidence of chronic hepatitis B infection will be allowed to enroll if on appropriate suppressive medications under the direction of a hepatologist and with PI approval
* Patients who are known to be positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) are not eligible
* Patients must not have live vaccine therapies for prevention of infectious diseases within 28 days of first nivolumab dose
* Patients who are unable to swallow oral medication are not eligible
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded; these include but are not limited to patients with a history of:

  * Immune related neurologic disease
  * Multiple sclerosis
  * Autoimmune (demyelinating) neuropathy
  * Guillain-Barre syndrome
  * Myasthenia gravis
  * Systemic autoimmune disease such as systemic lupus erythematosus (SLE)
  * Connective tissue diseases
  * Scleroderma
  * Inflammatory bowel disease (IBD)
  * Crohn's
  * Ulcerative colitis
  * Patients with a history of toxic epidermal necrolysis (TEN)
  * Stevens-Johnson syndrome
  * Anti-phospholipid syndrome NOTE: Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2017-08-27 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shira Dinner, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated for accrual on August 24, 2016 with the first patient enrolled and treated on the study on August 17, 2017. The study was terminated before the accrual goal of 22 patients was reached due to funding issues and slow accrual.
Period: Complete Cycle 1 (28 Days)
Arm/Group | Treatment (Dasatinib, Nivolumab)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Progressive disease/no response | 1
Period: Start Cycle 2 and Beyond
Arm/Group | Treatment (Dasatinib, Nivolumab)
Started | 0
Completed | 0
Not Completed | 0
Period: Follow-up for 1 Year
Arm/Group | Treatment (Dasatinib, Nivolumab)
Started (All patients that are treated on the study go into the follow-up period.) | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Dasatinib, Nivolumab)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-Limiting Toxicity (DLT)
Description: Determine the maximum tolerated dose (MTD) of nivolumab when given in combination with dasatinib, the MTD will be defined as the highest dose level at which ≤ 1 DLT occurs and will be assessed by the Common Terminology Criteria for Adverse Events version 4.03.
Time Frame: Up to 28 days
Population: Only one patient was treated on study and this patient did not complete the DLT period and was not evaluable for this outcome measure or any of the outcome measures. Sample size too small for analysis.
Arm/Group | Treatment (Dasatinib, Nivolumab)
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Adverse Events
Description: To evaluate the toxicity and safety of nivolumab and dasatinib in patients with relapsed/refractory Ph+ ALL. Adverse events will be assessed by number, frequency, and severity and will be graded according to the NCI's common terminology criteria, version 4.03.
Time Frame: Up to 28-days after the last dose
Reporting Status: Not Posted

3. Secondary Outcome: Rate of Complete Hematologic Remission (CR)
Description: Determine the rate of complete hematologic remission (CR) after three cycles of nivolumab and dasatinib
Time Frame: At 84 days (3 cycles)
Reporting Status: Not Posted

4. Secondary Outcome: Rate of Molecular Remission
Description: Determine the rate of molecular remission after three cycles of nivolumab and dasatinib.
Time Frame: At 84 days (3 cycles)
Reporting Status: Not Posted

5. Secondary Outcome: Serum Level of Dasatinib
Description: The serum level of dasatinib will be measured at 24 hours after the start of cycle 1 and on days 8, 15, and 22 prior to treatment during cycle 1.
Time Frame: 24 hours after the start of cycle 1 and days 8, 15, and 22 prior to treatment during cycle 1
Reporting Status: Not Posted

6. Secondary Outcome: Serum Level of Nivolumab
Description: The serum level of nivolumab will be measured on days 8, 15, and 22 prior to treatment during cycle 1.
Time Frame: Days 8, 15, and 22 prior to treatment during cycle 1
Reporting Status: Not Posted

7. Secondary Outcome: PD1 Expression Levels and Saturation Assessed in the Peripheral Blood
Description: Peripheral blood will be evaluated to measure PD1 expression levels and saturation.
Time Frame: Baseline to 28-days after the last dose
Reporting Status: Not Posted

8. Secondary Outcome: PD1 Expression Levels and Saturation in Bone Marrow
Description: Bone marrow will be assessed to measure PD1 expression levels and saturation.
Time Frame: Baseline to 28-days after the last dose
Reporting Status: Not Posted

9. Secondary Outcome: Peripheral T-cell Levels and Activation in Response to Treatment
Description: T-cell levels and activation will be measured in the peripheral blood after treatment.
Time Frame: At cycle 1 days: 1, 2, 8, 15, & 22 prior to dosing
Reporting Status: Not Posted

10. Other Pre Specified Outcome: The 30 Day Mortality Rate
Description: Number and percentage of patients that die within the first 30 days of initiating treatment.
Time Frame: Up to 30 days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Overall Survival (OS)
Description: OS is defined as the time from the initiation of study treatment until death from any cause, evaluated for up to 1 year.
Time Frame: Up to 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the initiation of study treatment until the time of disease progression or relapse.
Time Frame: Up to 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Duration of Remission (DOR)
Description: Duration of remission is defined as the time from achieving complete response until the time of disease relapse.
Time Frame: Up to 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Compare the OS Between Patients Who Receive a Hematopoietic Stem Cell Transplant and Those Who Receive no Further Therapy Following Remission
Time Frame: Up to 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Presence of Resistance Mutations in Bone Marrow at the Time of Disease Progression
Time Frame: Up to 28-days after the last dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The patient was monitored for AEs during treatment on the study and for 30 days after the last dose of study treatment (for approximately 40 days in duration).
Arm/Group | Treatment (Dasatinib, Nivolumab)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Dasatinib, Nivolumab) (N=1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Dasatinib, Nivolumab) (N=1)
Hyperglycemia (Metabolism and nutrition disorders) | 1
White blood cell decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Papulopustular rash (Infections and infestations) | 1
Hypertension (Vascular disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Hypotension (Vascular disorders) | 1
Lipase increased (Investigations) | 1
Sepsis (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lymphocyte count decreased (Investigations) | 1
INR increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Blood bilirubin increased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Anemia (Blood and lymphatic system disorders) | 1
Platelet count decreased (Investigations) | 1
Fatigue (General disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
The study was closed to accrual with only one patient enrolled. It did not meet its accrual goal of 22 patients due to slow accrual and funding issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT02819804/Prot_SAP_000.pdf